CLINICAL TRIAL: NCT02666547
Title: Value of PET/ CT in the 68Ga-NODAGA-RGD for the Evaluation of the Tumoral Neoangiogenesis
Brief Title: 68Ga-NODAGA-RGD PET/ CT for Tumoral Neoangiogenesis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of resources
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: George Coukos, MD PhD, Head of oncology (Unknown)
Responsible Party: Principal Investigator, John O. Prior, Chief Nuclear Medicine Department, University of Lausanne Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 220/12
Record Dates: First submitted 2016-01-24; First posted 2016-01-28 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Pathological Angiogenesis
Keywords: 68Ga-NODAGA-RGD; 18F-FDG; 18F-FET; PET/CT; neoangiogenesis
MeSH Terms: conditions — Neovascularization, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 68Ga-NODAGA-RGD,18F-FDG,18F-FET PET/CTs (Other): Active Comparator: 68Ga-NODAGA-RGD radiotracer All patients will undergo a 68Ga-NODAGA-RGD PET/CT, a 18F-FDG PET/CT or a 18F-FET PET/CT
  Interventions: Drug: 68Ga-NODAGA-RGD PET/CT; Radiation: 18F-FDG PET/CT; Radiation: 18F-FET PET/CT

INTERVENTIONS:
Drug: 68Ga-NODAGA-RGD PET/CT — 200 MBq 68 Ga-NODAGA-RGD will be administered i.v. and images acquired on all body . For glioma, images acquired centred on the skull
Radiation: 18F-FDG PET/CT — 3.5 MBq/kg 18F-FDG will be administered i.v. and images acquired on all body
Radiation: 18F-FET PET/CT — 200 MBq 18F-FET will be administered i.v. and images acquired centred on the skull

SUMMARY:
This study will assess the potential of the 68Ga-NODAGA-RGD for the evaluation of neoangiogenesis in patients followed for a neoplastic pathology and for whom a18F-FDG (or 18F-FET for gliomas) is indicated for initial extension evaluation or suspicion of recurrent tumor.

DETAILED DESCRIPTION:
The purpose of this study is to assess the value of 68Ga-NODAGA-RGD PET/CT for detection of neoangiogenesis at level of neoplastic processes, in patients, compared to 18F-FDG PET/CT (tumors other than glioma) or 18F-FET PET/CT (patients affected by glioma) and to determine the respective diagnostic contribution of every technique.

Every patient will undergo a routine 18F-FDG (or 18F-FET) PET/CT followed by a 68Ga-NODAGA-RGD PET / CT specific for the study within the next 7 days.

(each image procedure duration: 2h)

The criteria of primary evaluation for each of the techniques will be defined:

* On the images of PET/CT: SUVmax, SUVmoyen, VOI ( mL ), SUV41 % ratio [mean SUV of pixels ≥ 41 % of the SUVmax] of lesions / SUV
* On the images of CT: size of the lesions measured in 3D (axial, coronal and sagittal), density in Hounsfield unit (HU)

The 18F-FDG/18F-FET and 68Ga-NODAGA-RGD PET / CTs will be analyzed at first separately then will be compared according to the methods described in the analysis

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 85 years old
* Karnofsky index: ≥ 80%
* Patients presenting a neoplasic pathology, histologically proven, known to have expressed integrin αvβ3and for which a 18F-FDG (or a 18F-FETfor glioma) is indicated : (1) glioma (WHO I, II-IV), (2) malignant melanoma, (3) cancer of upper respiratory tract, (4) breast cancer,(5) bone metastasis, (6) ovarian cancer, (7) lung cancer,(8) non-Hodgkinian malignant lymphoma with extra- lymphatic nodes extension, (9) neuroendocrine tumors, (10) pancreatic cancer,(11) oesophagus cancer,(12) stomach cancer. 10 patients will be included per type of cancer.
* Informed consent signed

Exclusion Criteria:

* Incapacity to sign the informed consent
* Pregnancy, breastfeeding
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2023-08 (Actual); Study Completion 2023-09 (Actual)

PRIMARY OUTCOMES:
Comparison of each method of imaging for detection of tumors | within 10 days
  To compare the capacity of each of the techniques and their combination to detect tumors, to determine the composition of these tumors (neoangiogenesis, metabolism, necrosis), their extension, the changes due to treatment

SECONDARY OUTCOMES:
ROC analysis and comparison of areas under the curve | Within 10 days
  A ROC analysis will be realized as well as a comparison of AUCs, to determine the superiority of a method compared to the other one, using a parametric test comparing of the AUC curves and ROC curves respectively by an established algorithm. The criteria of interpretation and positivity will be defined in a standard way on the images 18F-FDG / 18F-FET and 68Ga-NODAGA-RGD.
Comparison 68Ga-NODAGA-RGD to standard routine extension imaging assessments | within 10 days
  The sensibility for detection of tumor by the 68Ga-NODAGA-RGD will be assessed and compared with the standard routine extension assessements including 18F-FDG PET/CT or18F-FET PET/CT, CT or any other complementary exam (US, MRI)

CONTACTS AND LOCATIONS:
Overall Officials: John O Prior, MD, PhD, Principal Investigator — Lausanne University Hospitals
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Nuclear Medicine, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Durante S, Dunet V, Gorostidi F, Mitsakis P, Schaefer N, Delage J, Prior JO. Head and neck tumors angiogenesis imaging with 68Ga-NODAGA-RGD in comparison to 18F-FDG PET/CT: a pilot study. EJNMMI Res. 2020 May 7;10(1):47. doi: 10.1186/s13550-020-00638-w. PMID 32382869
- [Derived] Dietz M, Dunet V, Mantziari S, Pomoni A, Dias Correia R, Testart Dardel N, Boughdad S, Nicod Lalonde M, Treglia G, Schafer M, Schaefer N, Prior JO. Comparison of integrin alphavbeta3 expression with 68Ga-NODAGA-RGD PET/CT and glucose metabolism with 18F-FDG PET/CT in esophageal or gastroesophageal junction cancers. Eur J Hybrid Imaging. 2023 Feb 1;7(1):3. doi: 10.1186/s41824-023-00162-9. PMID 36720731